CLINICAL TRIAL: NCT00122434
Title: A Randomized, Multiple-dose, Double-blind, Placebo- and Active-controlled, Parallel Group Efficacy and Safety Study to Determine the Optimum Dose of BEA 2180 BR Delivered by the Respimat® Inhaler in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Dose Finding Study in COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1205.4
Record Dates: First submitted 2005-07-18; First posted 2005-07-22 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

INTERVENTIONS:
Drug: BEA 2180 BR
Drug: tiotropium

SUMMARY:
The primary objective of this study is to determine the optimum dose of BEA 2180 BR inhalation solut ion delivered by the Respimat ? inhaler once daily for four weeks in patients with COPD.

ELIGIBILITY:
1. Patients must have relatively stable, moderate to severe airway obstruction with an FEV1 >=30% and <= 60% of predicted normal and FEV1 <=70% of FVC at the baseline PFTs at Visit 1 (at both timepoints).
2. All patients must have an increase in FEV1 of at least 12% from baseline (th e -10 minute measurement) 45 min after inhalation of 80 ?g Atrovent MDI.
3. Male or female patients 40 years of age or older.
4. Smoker or ex-smoker with a history of more than 10 pack years.

1. Patients with any other significant disease will be excluded. 2. Patients with a history of asthma or allergic rhinitis will be excluded.

Ages: 40 Years to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2005-07; Primary Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Trough forced expiratory volume (FEV1) response after four weeks of treatment. | 4 weeks

SECONDARY OUTCOMES:
Trough FEV1 response after 1 and 2 weeks | after 1 and 2 weeks
Trough FVC response after 1, 2 and 4 weeks | after 1, 2 and 4 weeks
FEV1, FVC AUC0-6h and peak response after 0, 1, 2 and 4 weeks | after 0, 1, 2 and 4 weeks
Individual FEV1 and FVC measurements at each time point | 4 weeks
Weekly mean pre-dose morning and evening PEFR | 4 weeks
Weekly mean number of occasions of rescue therapy used per day [as occasion requires (PRN) albuterol] | 4 weeks
COPD symptom scores (wheezing, shortness of breath, coughing and tightness of chest) | 4 weeks
Physician's Global Evaluation | 4 weeks
All adverse events | 7 weeks
Pulse rate and blood pressure (seated) recorded in conjunction with spirometry up to the three hour pulmonary function test (PFT) | 4 weeks
12-lead ECGs at baseline (-10 minutes) and at 25 minutes, 2 and 6 hours post dose (Visits 2 and 5) | 4 weeks
drug plasma concentrations | 4 or 7 weeks
drug urine concentrations | 4 or 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator
Locations (43):
- United States (27):
  - UAB Lung Health Center, Birmingham, Alabama
  - Vapahcs 111P, Palo Alto, California
  - Boehringer Ingelheim Investigational Site, San Diego, California
  - GLAHS Sepulveda, Sepulveda, California
  - Rehabilitation Clinical Trial Center, Torrance, California
  - Boehringer Ingelheim Investigational Site, Wheat Ridge, Colorado
  - Hospital for Special Care, New Britain, Connecticut
  - Bay Pines VA Medical Center, Bay Pines, Florida
  - Boehringer Ingelheim Investigational Site, Panama City, Florida
  - Boehringer Ingelheim Investigational Site, Pembroke Pines, Florida
  - Boehringer Ingelheim Investigational Site, Coeur d'Alene, Idaho
  - LSUHSC - Shreveport, Shreveport, Louisiana
  - VAMC-Reno, Reno, Nevada
  - North Shore Universtiy Hospital, New Hyde Park, New York
  - SVMMC, Toledo, Ohio
  - Boehringer Ingelheim Investigational Site, Medford, Oregon
  - Hershey Medical Center, Hershey, Pennsylvania
  - Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - Frank Sciurba, Pittsburgh, Pennsylvania
  - Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - MUSC, Charleston, South Carolina
  - Boehringer Ingelheim Investigational Site, Spartanburg, South Carolina
  - Boehringer Ingelheim Investigational Site, Harker Heights, Texas
  - MEDVAMC, Houston, Texas
  - McGuire VA, Fredericksburg, Virginia
  - Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - Boehringer Ingelheim Investigational Site, Tacoma, Washington
- Belgium (9):
  - CHU du Sart Tilman (B35), Angleur
  - A.Z. VUB, Brussels
  - UZ Antwerpen, Edegem
  - AZ Jan Palfijn, Ghent
  - UZ Gent, Ghent
  - Virga Jesseziekenhuis, Hasselt
  - Clinique Reine Astrid, Malmedy
  - Heilig Hartziekenhuis, Menen
  - Sint-Elisabethziekenhuis, Turnhout
- Netherlands (7):
  - Ziekenhuisgroep Twente, Almelo
  - Amphia Ziekenhuis, Breda
  - Tjongerschans Ziekenhuis, Heerenveen
  - Atrium Medisch Centrum, Heerlen
  - Ziekenhuisgroep Twente, Hengelo
  - Academisch Ziekenhuis Nijmegen St. Radbout, Nijmegen
  - Gelre Ziekenhuizen, Zutphen

REFERENCES:
- See also: Related Info — http://onlinelibrary.wiley.com/doi/10.1111/j.1440-1843.2012.02302.x/abstract